CLINICAL TRIAL: NCT03752801
Title: Improving Quality and Consistency in Family Education Prior to First Discharge Following Pediatric Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Pediatric Oncology Group of Ontario (Other)
Responsible Party: Principal Investigator, Denise Mills, Nurse Practitioner, The Hospital for Sick Children
Other Study IDs: REB1000060860
Record Dates: First submitted 2018-11-13; First posted 2018-11-26 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Oncology
Keywords: education; pediatric; family
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Script Review Parents/Caregivers: will have script reviewed and evaluated by parents/caregivers in groups of 5 up to 40 participants until 4/5 parents/caregivers demonstrate that script is understandable and acceptable.
- Video Review Parents/Caregivers: review and evaluation of the developed educational videos by parents/caregivers up to 20 parents who have not participated in the script review

SUMMARY:
When a child is diagnosed with cancer the family's world is turned upside down. Parents have high levels of stress because they must learn important information about their child's diagnosis,medications and treatments. They must also learn how to care for their child once they have left the safety of the hospital. Parents have voiced that during this time they receive too much information, have paper overload, and hear and read different information causing them to feel confused. Parents have shared that small amounts of information that can be repeated when they want and as often as they want helps them to feel more confident to care for their child. This study will ask parents if they like and can easily learn information about how to care for their child with cancer from short videos that highlight key points, have visual cues, and provide case examples. If parents find short videos useful and helpful for learning, with the goal that they will feel more confident to care for their child and have lower levels of anxiety.

DETAILED DESCRIPTION:
A diagnosis of childhood cancer is overwhelming for both the child and family. Parents/caregivers of newly diagnosed pediatric oncology patients need specialized education to provide safe care for their child at home. Previous research and clinical experience have highlighted that current strategies are not successful. Families report challenges with paper, information overload and teaching provided at a time when they are unable to focus. They describe inconsistent messages between different providers and sources of information.Parents/caregivers have expressed that information that is concise, consistent, with visual cues, and can be repeated, positively influences their ability to understand. Poor quality of discharge teaching in pediatrics is associated with increased emergency room visits and readmissions to hospital. Predictors of readmission include medical complexity and 4 or more medications prescribed at time of discharge. Pediatric oncology patients are medically complex and at risk for significant life-threatening complications. Multiple home medications are the standard for children receiving cancer therapy. Current parent/caregiver education is often driven by checklists of content that health careproviders (HCP) believe must be delivered prior to first hospital discharge. Timing of education is planned according to HCP schedules and not consistently at a time chosen by and suitable for parents/caregivers.

Methods for providing parent/caregiver education currently include verbal discussion with HCPs and written information. Evaluation of educational video strategies in pediatric oncology has been limited to taped diagnostic discussions. It is reported that 90% of parents/caregivers of pediatric cancer patients search the internet for information. Video education developed by pediatric oncology experts has the advantage of providing consistent information, being available for repeat viewing, and available at times chosen by the parents/caregivers.

Goals and Objectives The overarching goal is to improve consistency and quality of education provided to parents/caregivers of newly diagnosed pediatric oncology patients.

Primary Objective:

To develop two short video-based education modules for parents/caregivers of children with newly diagnosed cancer which are acceptable and understandable.

Secondary Objectives:

1. To determine the feasibility of a trial of providing education in video modules as demonstrated by the ability to recruit 20 parents/caregivers of newly diagnosed children with cancer within 8 months and by having at least 90% of enrolled parents/caregivers watch the two videos and answer 10 knowledge and confidence questions
2. To obtain qualitative feedback about the videos
3. To describe change in knowledge and confidence before and after viewing the two videos

Impact and Relevance Statement This study is proposing a novel video-based education program for parents/caregivers which hypothesize will lead to improved understanding and confidence to care for their child newly diagnosed with cancer post first discharge from hospital. Learning in this fashion can be conducted at a time best suited to each individual caregiver and allow for repetition of the materials as often as desired. It ensures that different caregivers for the same child receive the same information. The greatest impact will be on the parents/caregivers with a goal to increase knowledge, preparedness and confidence and minimize distress and anxiety.

Methods:

In this pilot study the investigators plan to develop and evaluate two video modules focused on two essential 'prior-to-first-discharge' topics: the approach to fever and giving medications at home. The video modules will be short, concise and will include case-based scenarios allowing parents/caregivers to review and consolidate teaching.

The content of the videos will be developed by pediatric oncology nurses, physicians and pharmacists from across POGO centers. The review panel will consist of 8-12 HCPs with representation by discipline and center. The script will be developed in a series of teleconferences in which first the content will be developed and refined using a consensus approach. Once the content is agreed upon, a script will be developed and refined among the review panel. When finalized, the investigators will begin to test acceptability and understandability with respondents. For this phase, eligible respondents will be any parent or caregiver of a child with cancer irrespective of type or timing of diagnosis. The investigators will exclude respondents who do not understand English. The investigators will then test the script with consecutive parent/guardian respondents using one-on-one cognitive interviews. The investigators will ask the respondent to read the script and the investigators will ask them to rate acceptability and understandability on 5 Point Likert scales which the investigators have used previously for instrument development.

Using a semi-structured interview, the investigators will ask probing questions to clarify their understanding of content. A second interviewer will be present who will rate understandability on a 4 point Likert scale ranging from 1=completely incorrect to 4=completely correct. After every 5 interviews, the results will be shared with the review panel who will decide whether to modify the script. Iterations will continue until at least 4 of the last 5 respondents are correct in their interpretation, state the script is understandable and acceptable and further modifications are not required based upon qualitative comments.

The finalized scripts will be developed into short videos, less than 5 minutes in length. The videos will be tested in new groups of 5 respondents and similarly evaluated for acceptability and understandability using cognitive interviews. Respondents will be specifically asked about length and clarity of information presented.

The videos will be considered satisfactory when at least 4 of the last 5 respondents are correct in their interpretation, state the video is understandable and acceptable and further modifications are not required based upon qualitative comments.

Confidence and knowledge questions will be developed in a similar method with consensus among the Pediatric Oncology HCPs and then with parents. This will allow both clinical expert consensus and parent validation.

Next, the investigators will test the feasibility of a trial of the educational video modules by conduct of a pilot study based at SickKids. Eligible respondents will be parents or caregivers of children newly diagnosed with cancer within the past 4 weeks. The investigators will exclude parents who do not understand English. Only one parent per child will be eligible. For eligible and consenting parents/caregivers, the investigators will ask them to watch the two videos, summarize the content of the video and provide feedback similar to the development phase. The investigators will also ask them to answer the confidence survey and the knowledge questions which will measure their knowledge and confidence in different domains of fever management and medication administration. The questions will be administered before and after watching the videos.

ELIGIBILITY:
Inclusion Criteria:

* for the first phase - review of script, eligible respondents will be any parent or caregiver of a child with cancer irrespective of type of timing of diagnosis.
* for the video review phase - must be a parent/caregiver of a child diagnosed with cancer in the last 8 months

Exclusion Criteria:

* must have written and spoken English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: parents or caregivers of children diagnosed with cancer
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Measure acceptability and ability to understand video-based education modules for parent/caregivers of children with newly diagnosed cancer | parents will watch video one (approx. 10 minutes)
  Develop 2 short video-based education modules for parents/caregivers of children with newly diagnosed cancer which are acceptable and understandable. This will be achieved when 90% of enrolled parents/caregivers watch the two videos and correctly answer 10 knowledge and confidence questions.

SECONDARY OUTCOMES:
Measure the feasibility of providing video to families | parents will watch video one (approx. 10 minutes)
  The feasibility of a trial of providing education in video modules as demonstrated by the ability to recruit 20 parents/caregivers of newly diagnosed children
Qualitative feedback about the videos | parents will watch video one (approx. 10 minutes)
  To obtain qualitative feedback about the videos. Qualitative feedback is being collected by asking the question "Is there anything else that you would like to tell us about the videos?"
Measure a change in knowledge and confidence before/after video | parents will watch video one (approx. 10 minutes) asked questions before the video and same questions at end of video
  To measure a change in knowledge and confidence before and after viewing the two videos. Scores on the knowledge and confidence questions will be compared before watching and after watching the videos.
  We utilized a likert scale to measure change with 1 = Not at all confident to 5= Extremely Confident

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mills, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Sickkids, Toronto, Ontario, Canada

REFERENCES:
- [Background] Landier W, Ahern J, Barakat LP, Bhatia S, Bingen KM, Bondurant PG, Cohn SL, Dobrozsi SK, Haugen M, Herring RA, Hooke MC, Martin M, Murphy K, Newman AR, Rodgers CC, Ruccione KS, Sullivan J, Weiss M, Withycombe J, Yasui L, Hockenberry M. Patient/Family Education for Newly Diagnosed Pediatric Oncology Patients. J Pediatr Oncol Nurs. 2016 Nov/Dec;33(6):422-431. doi: 10.1177/1043454216655983. Epub 2016 Jul 9. PMID 27385664
- [Background] Haugen MS, Landier W, Mandrell BN, Sullivan J, Schwartz C, Skeens MA, Hockenberry M. Educating Families of Children Newly Diagnosed With Cancer. J Pediatr Oncol Nurs. 2016 Nov/Dec;33(6):405-413. doi: 10.1177/1043454216652856. Epub 2016 Jul 8. PMID 27268501
- [Background] Rodgers CC, Laing CM, Herring RA, Tena N, Leonardelli A, Hockenberry M, Hendricks-Ferguson V. Understanding Effective Delivery of Patient and Family Education in Pediatric OncologyA Systematic Review From the Children's Oncology Group [Formula: see text]. J Pediatr Oncol Nurs. 2016 Nov/Dec;33(6):432-446. doi: 10.1177/1043454216659449. Epub 2016 Jul 27. PMID 27450361
- [Background] Rodgers CC, Stegenga K, Withycombe JS, Sachse K, Kelly KP. Processing Information After a Child's Cancer Diagnosis-How Parents Learn. J Pediatr Oncol Nurs. 2016 Nov/Dec;33(6):447-459. doi: 10.1177/1043454216668825. PMID 28084180
- [Background] Weiss ME, Costa LL, Yakusheva O, Bobay KL. Validation of patient and nurse short forms of the Readiness for Hospital Discharge Scale and their relationship to return to the hospital. Health Serv Res. 2014 Feb;49(1):304-17. doi: 10.1111/1475-6773.12092. Epub 2013 Jul 16. PMID 23855675
- [Background] O'Sullivan C, Dupuis LL, Gibson P, Johnston DL, Baggott C, Portwine C, Spiegler B, Kuczynski S, Tomlinson D, de Mol Van Otterloo S, Tomlinson GA, Sung L. Refinement of the symptom screening in pediatrics tool (SSPedi). Br J Cancer. 2014 Sep 23;111(7):1262-8. doi: 10.1038/bjc.2014.445. Epub 2014 Aug 7. PMID 25101569